CLINICAL TRIAL: NCT05579951
Title: Randomised Control Trial of Patient Specific Instrumentation vs Standard Instrumentation of the GMK-Sphere (Global Medacta Knee) Total Knee Arthroplasty
Brief Title: Bespoke vs Standard Instrumentation in TKR
Acronym: SPHERE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R04611
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty; Stability; Osteoarthritis; Knee; Functional Outcome; Gait; Patient Specific Instrumentation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Total knee replacement with conventional instrumentation
  Interventions: Procedure: Conventional
- Patient specific instrumentation (Active Comparator): Total knee replacement with patient specific instrumentation
  Interventions: Procedure: Patient specific instrumentation; Device: Patient specific instrumentation

INTERVENTIONS:
Procedure: Patient specific instrumentation — Total knee replacement with patient specific instrumentation
  Arms: Patient specific instrumentation
Procedure: Conventional — Total knee replacement with conventional instrumentation
  Arms: Conventional
Device: Patient specific instrumentation — Medacta GMK Sphere MyKnee Patient specific Instrumentation
  Arms: Patient specific instrumentation

SUMMARY:
Total knee replacements are operations that are offered to patients who have severe arthritis pain that is affecting daily activities that is no longer controlled with painkillers. The operation will replace the worn joints with metal implants and a plastic spacer. Total knee replacements are successful operations in the vast majority of patients. However, a small minority of patients are not entirely satisfied with the outcome of their knee replacement. Researchers are studying whether the precise positioning of the implant has an effect on the outcome.

This study will look at whether patient-specific instrumentation improves implant position and if it leads to improved patient function so that we know what to recommend in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis of the knee which is sufficiently symptomatic to require knee arthroplasty as assessed by their consultant orthopaedic surgeon

Exclusion Criteria:

* Patients with inflammatory arthropathy, patients requiring bone augmentation, patients with ligament incompetence or valgus deformity >5 degrees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Gait Kinematics at 1-Year | 1 year post-operatively
  Gait of patients will be analysed pre-operatively, six-weeks post-operatively, and 1-year post-operatively by 3D motion capture technology. The change measured over time at 1-year will be the primary outcome.

SECONDARY OUTCOMES:
Patient Satisfaction (Pain/Hospital experience/functional ability/Surgery expectations) | 1 year post-operatively
  Patient satisfaction will be reported using a scale on a questionnaire which asks six questions on how happy patients were with their hospital experience/level of pain/functional ability post-operatively. The questionnaire also asks whether their expectations were met. The two satisfaction questions are answered on a scale of 'Very Satisfied/Satisfied/Unsure/Dissatisfied' by ticking the appropriate box. The four questions based on patient expectation are scored on a scale of 'Excellent/Good/Unsure/Poor' by ticking the appropriate box.
Oxford Knee Score (Patient reported outcome measure of pain and function) | 6 weeks post-operatively
  A joint specific questionnaire which asks patients on the level of pain and function they believe to have in their affected knee (taking into consideration the past 4 weeks only). The questionnaire consists of 12 questions. Five of the questions are pain related, and seven are aimed at function. Each question has 5 options and is scored from 0-4, with 4 being the best and 0 being the worst pain/function. The best score is therefore 48 (no pain/good function), and the worst score is 0 (pain and poor function).
Oxford Knee Score (Patient reported outcome measure of pain and function) | 1 year post-operatively
  A joint specific questionnaire which asks patients on the level of pain and function they believe to have in their affected knee (taking into consideration the past 4 weeks only). The questionnaire consists of 12 questions. Five of the questions are pain related, and seven are aimed at function. Each question has 5 options and is scored from 0-4, with 4 being the best and 0 being the worst pain/function. The best score is therefore 48 (no pain/good function), and the worst score is 0 (pain and poor function).
EuroQol-5 Dimensions (EQ-5D) (Patient reported outcome measure of patients' perception of their overall health) | 6 weeks post-operatively
  A questionnaire on patients' perception of their overall health. The questionnaire focuses on generic health in 5 dimensions: Mobility, self-care, pain or discomfort, anxiety or depression and usual activities (including work, housework, leisure, family, and study). The questions are scored using an algorithm; the result of which relates to the health status of the patient. This score ranges between 0 (equivalent to death) to 1 (equivalent to full health). It also contains a visual analogue scale where patients have to choose on a scale of 0-100 how well they believe their general health to be on that particular day, where 0 is the worst health imaginable and 100 is the best health imaginable.
EuroQol-5 Dimensions (EQ-5D) (Patient reported outcome measure of patients' | 1 year post-operatively
  A questionnaire on patients' perception of their overall health. The questionnaire focuses on generic health in 5 dimensions: Mobility, self-care, pain or discomfort, anxiety or depression and usual activities (including work, housework, leisure, family, and study). The questions are scored using an algorithm; the result of which relates to the health status of the patient. This score ranges between 0 (equivalent to death) to 1 (equivalent to full health). It also contains a visual analogue scale where patients have to choose on a scale of 0-100 how well they believe their general health to be on that particular day, where 0 is the worst health imaginable and 100 is the best health imaginable.
Short Form-12 (SF-12) (Patient reported outcome measure of general quality of life) | 6 weeks post-operatively
  A general Quality of Life score with 12 questions. It has mental and physical components which are scored from the same questions, using different algorithms. Each question is multiple choice, and the patient must tick one answer. Each answer corresponds to a standardised value, which is used in two algorithms to generate an overall score. One score is for the mental component and one is for the physical component. The physical standardized values are summed across all 12 items. 56.57706 is added to the sum to create the SF-12 physical score. 60.75781 is added to sum create the SF-12 mental score. Higher overall scores are better than lower scores.
Short Form-12 (SF-12) (Patient reported outcome measure of general quality of life) | 1 year post-operatively
  A general Quality of Life score with 12 questions. It has mental and physical components which are scored from the same questions, using different algorithms. Each question is multiple choice, and the patient must tick one answer. Each answer corresponds to a standardised value, which is used in two algorithms to generate an overall score. One score is for the mental component and one is for the physical component. The physical standardized values are summed across all 12 items. 56.57706 is added to the sum to create the SF-12 physical score. 60.75781 is added to sum create the SF-12 mental score. Higher overall scores are better than lower scores.
Knee range of motion | 6 weeks post-operatively
  Knee range of motion in degrees will be assessed using a goniometer
Knee range of motion | 1 year post-operatively
  Knee range of motion in degrees will be assessed using a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Leela Biant, Principal Investigator — University of Manchester
Locations (1):
- Trafford General Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Study protocol and participant facing documents can be shared to other researchers upon request to the research team. Requests can be emailed to MORE@manchester.ac.uk